CLINICAL TRIAL: NCT04929873
Title: Clinical Study of VA-ECMO Remote Limb Re-perfusion Monitoring Technology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-567
Record Dates: First submitted 2021-06-01; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-05

CONDITIONS: Perfusion; Complications

STUDY DESIGN:
Intervention Model Description: transdynation for real-time pressure monitoring
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- routine treatment (Placebo Comparator): routine nursing
  Interventions: Behavioral: Routine monitor
- Experimental group (Experimental): Immediately after the establishment of the side branch cycle, the closed transdone is connected for real-time monitoring of pressure, and clinical nursing practice is guided by transdictor pressure.
  Interventions: Behavioral: Closed transdyser

INTERVENTIONS:
Behavioral: Closed transdyser — When the average arterial pressure ≥ 50mmHg, it is indicated that the basic blood supply of the lower extremities is satisfied without special treatment, and when the average arterial pressure < 50mmHg, it indicates insufficient perfusion, by adjusting the pipe position, changing the ECMO flow rate, and properly clamping the artery end to divert part of the blood flow to the side branch circulation, so that the average arterial pressure is maintained above 50mmHg.
  Arms: Experimental group
Behavioral: Routine monitor — Obtain oxygen saturation, skin color, temperature, etc
  Arms: routine treatment

SUMMARY:
Establish and verify the feasibility and effectiveness of VA-ECMO remote limb re-perfusion monitoring technology.

DETAILED DESCRIPTION:
It is proposed to monitor VA-ECMO arterial end side branch circulation in real time through a set of monitoring equipment, guide clinical adjustment, improve lower limb re-perfusion, reduce the occurrence of lower limb ischemia, in order to achieve the goal of early detection, early prevention and early treatment, and provide reference and theoretical basis for clinical practice.

Monitoring techniques are divided into two parts: A. monitoring equipment (connecting transdiotic monitoring pressure on va-ECMO side branches cycle); B.to guide clinical adjustment by monitoring pressure (average arterial pressure).

ELIGIBILITY:
Inclusion Criteria:

* Age: adult patients ≥ 18 years of age;
* signed ECMO informed consent;
* femur vein VA-ECMO treatment;
* agreed to establish VA-ECMO side branch cycle;
* informed consent to this study.

Exclusion Criteria:

* a completely closed double lower limb venously before surgery;
* amputee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of ischemia Incidence of ischemia | 1 year
  of ischemia in the lower extremities on the side of the tube

CONTACTS AND LOCATIONS:
Overall Officials: Fei Zeng, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- SAHZhejiangU, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No